CLINICAL TRIAL: NCT07367334
Title: Impact of Verbal Cueing in Multimodal Exercise Rehabilitation: A Retrospective Study in Breast Cancer Survivors Undergoing Radiation Therapy
Brief Title: Effects of MMV Exercise With and Without Verbal Guidance on Shoulder Movement, Fatigue, and Stress in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saveetha University (Other)
Responsible Party: Principal Investigator, Tamil Ponni Sivamani, Principal Investigator, Saveetha University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 064/05/2025/ISRB/PGSR/SCPT
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Survivors; Range of Motion; Cortisol; Shoulder Dysfunction; Fatigue After Adjuvant Breast Cancer Treatment
Keywords: Good Health and Well-Being; Quality Education; Quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodel Exercise with Verbal cues (Experimental)
  Interventions: Other: Multimodal Exercise Rehabilitation With Verbal Cueing
- Multimodel Exercise without Verbal cues (Active Comparator)
  Interventions: Other: Multimodel Exercises Rehabilitation without Verbal cues

INTERVENTIONS:
Other: Multimodal Exercise Rehabilitation With Verbal Cueing — The intervention consisted supervised multimodal exercise rehabilitation program designed for breast cancer survivors undergoing radiation therapy. Each exercise session lasted approximately 45 minutes and includes aerobic exercises, resistance training, flexibility exercises, and relaxation techniques aimed at improving shoulder mobility, reducing cancer-related fatigue, and regulating physiological stress. The program is delivered three times per week for 12 weeks, with exercise intensity and progression tailored to individual tolerance and safety. In one arm, exercises are delivered with structured verbal cueing provided by the therapist, including instructions, corrective feedback, breathing guidance, pacing, and motivational support throughout the session. In the comparison arm, the same exercises are performed without verbal cueing after an initial demonstration.
  Arms: Multimodel Exercise with Verbal cues
Other: Multimodel Exercises Rehabilitation without Verbal cues — Participants in this arm received a supervised multimodal exercise rehabilitation program conducted without verbal cueing. Each exercise session lasted approximately 45 minutes and is performed three times per week for 12 weeks. The program includes aerobic exercises, resistance training, flexibility exercises, and relaxation techniques aimed at improving shoulder mobility, reducing cancer-related fatigue, and regulating physiological stress.
  Participants performed the exercises following an initial demonstration, without ongoing verbal instructions, feedback, or encouragement during exercise execution. Exercise frequency, duration, intensity, and progression are standardized and identical to the verbal cueing group, ensuring consistency across interventions. The absence of verbal cueing allows evaluation of the effects of exercise delivery without therapist-guided verbal input.
  Arms: Multimodel Exercise without Verbal cues

SUMMARY:
The goal of this clinical trial is to learn whether a multimodal exercise rehabilitation program with verbal cueing is more effective than the same exercise program without verbal cueing in improving shoulder movement, reducing fatigue, and lowering stress levels in adult female breast cancer survivors undergoing radiation therapy.

The main questions it aims to answer are:

Does a multimodal exercise program with verbal cues improve shoulder range of motion more than the same program without verbal cues? Does verbal cueing during exercise reduce cancer-related fatigue more effectively than exercise without verbal cues? Does verbal cue-based exercise lead to greater improvement in salivary cortisol levels compared to exercise without verbal cues?

Researchers will compare multimodal exercise with verbal cues to multimodal exercise without verbal cues to see if verbal guidance improves physical function, fatigue, and stress regulation.

Participants will be adult female breast cancer survivors undergoing radiation therapy who are enrolled in this clinical trial. Eligible participants will be assigned to one of two groups and will take part in a supervised multimodal exercise rehabilitation program for a duration of 12 weeks. Depending on group allocation, participants will perform the same set of exercises either with structured verbal cues provided by the therapist or without verbal cues. Throughout the study period, participants will attend regular exercise sessions and follow the prescribed exercise protocol. Shoulder range of motion will be assessed using standard goniometric measurements, cancer-related fatigue will be evaluated using the FACIT-Fatigue questionnaire, and physiological stress will be measured through salivary cortisol levels. All assessments will be conducted before the start of the exercise program and again at the end of the 12-week intervention period.

DETAILED DESCRIPTION:
Breast cancer survivors undergoing radiation therapy frequently experience shoulder dysfunction, cancer-related fatigue, and increased physiological stress, which adversely affect functional ability and quality of life. Exercise-based rehabilitation is known to improve physical and psychological outcomes in this population; however, the added value of verbal cueing during exercise has not been clearly established.

This clinical trial evaluates the effectiveness of a multimodal exercise rehabilitation program delivered with verbal cues compared to the same program delivered without verbal cues. The multimodal exercise program includes aerobic training, resistance exercises, flexibility exercises, and relaxation techniques aimed at improving shoulder mobility, reducing fatigue, and regulating stress responses. Verbal cueing involves therapist-provided instructions, feedback, and encouragement intended to enhance motor learning, exercise execution, and participant engagement.

Participants are assigned to one of two groups and complete a supervised 12-week exercise program. Both groups follow identical exercise protocols in terms of frequency, duration, and intensity, differing only in the presence or absence of verbal guidance. Outcomes are assessed at baseline and post-intervention. Shoulder range of motion is measured using goniometry, fatigue is evaluated using the FACIT-Fatigue scale, and physiological stress is assessed through salivary cortisol levels.

This study aims to determine whether verbal cueing enhances the effectiveness of multimodal exercise rehabilitation and to support evidence-based physiotherapy strategies for improving functional recovery and well-being in breast cancer survivors undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria: •Female breast cancer survivors (≥3 months, ≤5 years' post-diagnosis)

* Age group: 35-45 years
* FACIT-Fatigue score ≤ 34
* Salivary cortisol levels: 15-30 ng/mL (morning range)
* ROM minimum of 50% of the normal range of motion in the affected shoulder, specifically in the movements of flexion, abduction, and external rotation.

Exclusion Criteria: •Active infection or severe Graft vs Host Disease (GVHD)

* Psychiatric or cognitive impairments
* Severe comorbidities
* Inability to participate in exercise
* Severe fatigue
* Electrolyte imbalance
* Acute organ dysfunction (liver/kidney/lung)
* Active bleeding or recent surgery
* Recent transplantation (e.g., stem cell therapy)

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of motion | 12 weeks (Base line and 12th Week)
  Shoulder range of motion was assessed as a primary functional outcome, focusing on shoulder flexion, abduction, and external rotation of the affected upper limb. Active ROM was measured using a standard universal goniometer following standardized anatomical landmarks and testing positions. Assessments were performed at baseline and after completion of the intervention period. Improvements in shoulder ROM indicate enhanced joint mobility, soft tissue flexibility, and functional use of the upper limb. Goniometric measurement is a reliable and widely accepted method for evaluating shoulder function in oncological rehabilitation.

SECONDARY OUTCOMES:
FACIT-Fatigue Scale | 12 Weeks (Baseline and 12th week)
  Cancer-related fatigue was evaluated using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale, a validated, self-administered questionnaire designed specifically to assess fatigue and its impact on daily functioning in individuals with chronic illness, including cancer. The FACIT-F consists of 13 items rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("very much"), with total scores ranging from 0 to 52. Higher scores indicate lower levels of fatigue and better functional well-being. Participants completed the questionnaire at baseline and following the completion of the intervention period. Fatigue is one of the most prevalent and persistent symptoms experienced by breast cancer survivors undergoing radiation therapy and can significantly impair physical performance, emotional health, and quality of life. The FACIT-F Scale has demonstrated excellent reliability, validity, and sensitivity to change in oncology population
Salivary Cortisol Level | 12 Weeks (Baseline and 12th Week)
  Physiological stress response was assessed through the measurement of salivary cortisol levels, a non-invasive biomarker reflecting hypothalamic pituitary adrenal (HPA) axis activity. Saliva samples were collected under standardized conditions to minimize the influence of diurnal variation in cortisol secretion. Samples were obtained at consistent times of the day both before and after the intervention period. Elevated cortisol levels are commonly associated with chronic stress, fatigue, and disrupted neuroendocrine regulation in breast cancer survivors undergoing active treatment. A reduction or normalization of salivary cortisol levels following the intervention indicates improved stress regulation, enhanced autonomic balance, and better physiological adaptation to treatment-related stress.

CONTACTS AND LOCATIONS:
Overall Officials: Shenbaga Sundaram Subramanian, Principal Investigator — Saveetha College of Physiotherapy, Saveetha Institute of medical and technical sciences (SIMATS)
Locations (1):
- Saveetha Medical College and hospital (SMCH), Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guardamagna L, Diamanti O, Artioli G, Casole L, Bernardi M, Bonadies F, Zennaro E, Modena GM, Nania T, Dellafiore F. Breast Cancer Survivors' Perception on Health Promotion and Healthy Lifestyle: A Systematic Review and Qualitative Meta-Synthesis. Int J Environ Res Public Health. 2025 Jul 17;22(7):1131. doi: 10.3390/ijerph22071131. PMID 40724197
- [Result] Gupta B, Gupta K, Narula K, Sharma P, Mittal A. The Effect of Exercise on Quality of Life among Patients and Survivors of Breast Cancer: A Systematic Review and Meta-Analysis. Asian Pac J Cancer Prev. 2025 Mar 1;26(3):715-723. doi: 10.31557/APJCP.2025.26.3.715. PMID 40156386
- [Result] Zhang Y, Ji Y, Liu S, Li J, Wu J, Jin Q, Liu X, Duan H, Feng Z, Liu Y, Zhang Y, Lyu Z, Song F, Song F, Yang L, Liu H, Huang Y. Global burden of female breast cancer: new estimates in 2022, temporal trend and future projections up to 2050 based on the latest release from GLOBOCAN. J Natl Cancer Cent. 2025 Feb 13;5(3):287-296. doi: 10.1016/j.jncc.2025.02.002. eCollection 2025 Jun. PMID 40693239
- [Result] Xiong X, Zheng LW, Ding Y, Chen YF, Cai YW, Wang LP, Huang L, Liu CC, Shao ZM, Yu KD. Breast cancer: pathogenesis and treatments. Signal Transduct Target Ther. 2025 Feb 19;10(1):49. doi: 10.1038/s41392-024-02108-4. PMID 39966355

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT07367334/Prot_SAP_ICF_000.pdf